CLINICAL TRIAL: NCT05564117
Title: Efficacy and Safety of Oral Semaglutide 25 mg Once Daily in Adults With Overweight or Obesity
Brief Title: Research Study Looking at How Well Semaglutide Tablets Taken Once Daily Work in People Who Have a Body Weight Above the Healthy Range
Acronym: OASIS 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9932-4954; U1111-1271-9056 (Other: World Health Organization (WHO)); 2021-006534-40 (EudraCT Number)
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral semaglutide 25 mg (Experimental): Participants will receive semaglutide tablets orally once daily. Participants will receive semaglutide in a dose escalation manner for 64 weeks: 3 mg (weeks 0 to 4), 7 mg (weeks 5 to 8), 14 mg (weeks 9 to 12), and 25 mg (weeks 13 to 64).
  Interventions: Drug: Semaglutide
- Oral semaglutide placebo (Placebo Comparator): Participants will receive placebo tablets matched to semaglutide orally once daily for 64 weeks.
  Interventions: Drug: Placebo semaglutide

INTERVENTIONS:
Drug: Semaglutide — Semaglutide tablets orally once daily for 64 weeks.
  Arms: Oral semaglutide 25 mg
Drug: Placebo semaglutide — Semaglutide placebo-matching tablets orally once daily for 64 weeks.
  Arms: Oral semaglutide placebo

SUMMARY:
This study will look how well semaglutide tablets taken once daily helps people with body weight above the healthy range. Participants will either get semaglutide 25 milligram (mg) once daily or placebo once daily. This study will last for 72 weeks, which includes 1-week screening period, 64 weeks of treatment period and 7 weeks of follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study
* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Body mass index (BMI) of
* Greater than or equal to 27.0 kg/m^2 with the presence of at least one of the following weight-related complications (treated or untreated): hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular (CV) disease OR
* Greater than or equal to 30.0 kg/m^2
* History of at least one self-reported unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* A self-reported change in body weight greater than 5 kg (11 pound [lbs]) within 90 days before screening irrespective of medical records
* HbA1c greater than or equal to 6.5 percent (48 mmol/mol) as measured by the central laboratory at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 64)
  Measured in percentage (%).
Number of participants who achieve body weight loss equal to or above 5 percent (yes/no) | At end of treatment (week 64)
  Measured as count of participants.

SECONDARY OUTCOMES:
Number of participants who achieve body weight loss equal to or above 10 percent (yes/no) | At end of treatment (week 64)
  Measured as count of participants.
Number of participants who achieve body weight loss equal to or above 15 percent (yes/no) | At end of treatment (week 64)
  Measured as count of participants.
Number of participants who achieve body weight loss equal to or above 20 percent (yes/no) | At end of treatment (week 64)
  Measured as count of participants.
Change in Impact of Weight on Quality of Life-Lite-Clinical Trials version (IWQOL-Lite-CT) (Physical Function Domain [5-items] Score) | From baseline (week 0) to end of treatment (week 64)
  The Impact of Weight on Quality of Life Clinical Trials Version (IWQOL-Lite-CT) is designed to assess the impact of changes in weight on participant's quality of life within the context of clinical trials. IWQOL-Lite-CT is a 20-item questionnaire-based instrument used to assess the impact of body weight changes on participant's overall health-related quality of life (HRQoL). All IWQOL-Lite-CT composite scores range from 0 to 100, with higher scores reflecting better levels of functioning.
Change in body mass index (BMI) | From baseline (week 0) to end of treatment (week 64)
  Measured in kilogram per square meter (kg/m^2).
Change in waist circumference | From baseline (week 0) to end of treatment (week 64)
  Measured in centimeter (cm).
Change in systolic blood pressure | From baseline (week 0) to end of treatment (week 64)
  Measured in millimeter of mercury (mmHg).
Change in diastolic blood pressure | From randomisation (week 0) to end of treatment (week 64)
  Measured in mmHg.
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 64)
  Measured in percentage point (%-point).
Change in lipid: Total cholesterol (ratio to baseline) | From baseline (week 0) to end of treatment (week 64)
  Change from baseline in total cholesterol at week 64 will be presented as ratio to baseline.
Change in lipid: High-density lipoprotein (HDL) cholesterol (ratio to baseline) | From baseline (week 0) to end of treatment (week 64)
  Change from baseline in HDL cholesterol at week 64 will be presented as ratio to baseline.
Change in lipid: Low-density lipoprotein (LDL) cholesterol (ratio to baseline) | From baseline (week 0) to end of treatment (week 64)
  Change from baseline in LDL cholesterol at week 64 will be presented as ratio to baseline.
Change in lipid: Very-low-density lipoprotein (VLDL) cholesterol (ratio to baseline) | From baseline (week 0) to end of treatment (week 64)
  Change from baseline in VLDL cholesterol at week 64 will be presented as ratio to baseline.
Change in lipid: Triglycerides (ratio to baseline) | From baseline (week 0) to end of treatment (week 64)
  Change from baseline in triglycerides at week 64 will be presented as ratio to baseline.
Change in lipid: Free fatty acids (ratio to baseline) | From baseline (week 0) to end of treatment (week 64)
  Change from baseline in free fatty acids at week 64 will be presented as ratio to baseline.
Change in high sensitivity C Reactive Protein | From baseline (week 0) to end of treatment (week 64)
  Change from baseline in high sensitivity C Reactive Protein at week 64 will be presented as ratio to baseline.
Change in fasting plasma glucose (FPG) | From baseline (week 0) to end of treatment (week 64)
  Change from baseline in FPG at week 64 will be presented as ratio to baseline.
Change in fasting serum insulin | From baseline (week 0) to end of treatment (week 64)
  Change from baseline in fasting serum insulin at week 64 will be presented as ratio to baseline.
Number of treatment emergent adverse events | From baseline (week 0) to end of study (week 71)
  Measured as count of events.
Number of treatment emergent serious adverse events | From baseline (week 0) to end of study (week 71)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (23):
- United States (7):
  - Univsty Of AL At Birmingham, Birmingham, Alabama
  - FDRC, Costa Mesa, California
  - East West Medical Research Institute_Honolulu, Honolulu, Hawaii
  - Accellacare, Wilmington, North Carolina
  - UT Southwestern Med Cntr, Dallas, Texas
  - Washington Cntr Weight Mgmt, Arlington, Virginia
  - Selma Medical Associates, Winchester, Virginia
- Canada (2):
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Wharton Med Clin Trials, Hamilton, Ontario
- Germany (8):
  - InnoDiab Forschung GmbH, Essen
  - Diabetologische Gemeinschaftspraxis Dr. Staudenmeyer und Dr. Schiwietz, Lingen
  - MedicalCenter am Clemenshospital - Schwerpunktpraxis für Diabetologie und Ernährungsmedizin, Münster
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Praxis Dr. med. Wenzl-Bauer, Rehlingen-Siersburg
  - MZM Praxis Drs. Erlinger, Stuttgart
  - Jacob, Villingen-Schwenningen, Villingen-Schwenningen
  - Zentrum für klinische Studien Allgäu Oberschwaben, Wangen
- Poland (6):
  - Beata Miklaszewicz&Dariusz Dabrowski "CARDIAMED" s.j., Legnica, Lower Silesian Voivodeship
  - ETG Lublin, Lublin, Lublin Voivodeship
  - ETG Siedlce, Siedlce, Masovian Voivodeship
  - ETG Warszawa Sp. z o.o., Warsaw, Masovian Voivodeship
  - Gabinet Leczenia Otylosci i Chorob Dietozaleznych, Bialystok, Podlaskie Voivodeship
  - Centrum Zdrowia Metabolicznego, Poznan, Wielkopolskie Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.

REFERENCES:
- [Derived] Wharton S, Lingvay I, Bogdanski P, Duque do Vale R, Jacob S, Karlsson T, Shaji C, Rubino D, Garvey WT; OASIS 4 Study Group. Oral Semaglutide at a Dose of 25 mg in Adults with Overweight or Obesity. N Engl J Med. 2025 Sep 18;393(11):1077-1087. doi: 10.1056/NEJMoa2500969. PMID 40934115